CLINICAL TRIAL: NCT02072044
Title: A Phase II Study of Anlotinib(AL3818) in Patients With Advanced Renal Cell Carcinoma(RCC) That Have Failed Or Are Intolerant To TKIs Therapy
Brief Title: Phase II Study of Anlotinib in Patients With Advanced Renal Cell Carcinoma That Have Failed Or Are Intolerant To TKIs Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-06-IIB
Record Dates: First submitted 2014-01-20; First posted 2014-02-26 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma（RCC）; Anlotinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — anlotinib

ARMS (1):
- Anlotinib (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd

SUMMARY:
Anlotibib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2、VEGFR3、PDGFRβ and c-Kit. It has the obvious resistance to new angiogenesis. The trial is to explore the efficacy and safety profile of Anlotinib in patients with advanced Renal Cell Carcinoma(RCC) that have failed to TKIs therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with histologically confirmed advanced renal cell carcinoma including clear cell component and not available for surgery
* 2.Previously Failed Or Are Intolerant To TKIs Therapy(such as sunitinib, Sorafenib)
* 3.With measurable disease (using RECIST1.1)
* 4.18-75years,ECOG PS:0-1,Life expectancy of more than 3 months
* 5.Last TKIs Therapy≥4 weeks
* 6.Main organs function is normal
* 7.Signed and dated informed consent

Exclusion Criteria:

* 1.patients has many influence factors toward oral medications
* 2.Known brain metastases
* 3.patients with severe and failed to controlled diseases,including: suboptimal blood pressure control;suffering from myocardial ischemia or above grade I myocardial infarction, arrhythmias and Class I heart failure;activity or failure to control severe infections;liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis;poorly controlled diabetes (FBG)>10mmol/L);urine protein≥++,etc.
* 4.patients failed to heal wounds or fractures for Long-term
* 5.patients occurred venous thromboembolic events within 6 months
* 6.patients has HIV-positive or organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | each 42 days up to PD or death (up to 36 months)
  The PFS time is defined as time from randomization to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of: "death", "last tumor assessment", "last follow up date" or "last date in drug log"

SECONDARY OUTCOMES:
Objective Response Rate | each 42 days up to intolerance the toxicity or PD (up to 36 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule by enhanced CT/MRI scan every two cycles. Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 36 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule by enhanced CT/MRI scan every two cycles. Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
Overall Survival (OS) | From randomization until death (up to 36 months)
  OS was defined as time from date of randomization to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi medical university affiliated tumor hospital, Nanning, Guangxi
  - Harbin medical university affiliated tumor hospital, Haerbin, Heilongjiang
  - The 81st Hospital of Chinese PLA, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - China General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Qilu Hospital，Shandong University, Jinan, Shandong
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Ma J, Song Y, Shou J, Bai Y, Li H, Xie X, Luo H, Ren X, Liu J, Ye D, Bai X, Fu C, Qin S, Wang J, Zhou AP. Anlotinib for Patients With Metastatic Renal Cell Carcinoma Previously Treated With One Vascular Endothelial Growth Factor Receptor-Tyrosine Kinase Inhibitor: A Phase 2 Trial. Front Oncol. 2020 May 7;10:664. doi: 10.3389/fonc.2020.00664. eCollection 2020. PMID 32457838
- See also: Cancer — http://clinicaltrials.gov/ct2/bye/uQoPWw4lZX-i-iSxudhWudNzlXNiZip9m67PvQ7xzwhaLwS90B7x061nuQoPmdt.
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp